CLINICAL TRIAL: NCT01800604
Title: Psychological Treatment of Disability-Related Pain: Efficacy and Mechanisms
Brief Title: Power Over Pain (POP) Study
Acronym: POP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Washington (Other)
Collaborators: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH); National Institutes of Health (NIH) (NIH)
Responsible Party: Principal Investigator, Mark Jensen, Professor, Rehabilitative Medicine, University of Washington
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 43605; 1R01HD070973 (NIH)
Record Dates: First submitted 2013-02-08; First posted 2013-02-27 (Estimated); Last update posted 2018-10-17 (Actual); Status verified 2018-10

CONDITIONS: Multiple Sclerosis; Spinal Cord Injury; Chronic Pain; Other and Unspecified Amputation Stump Complications; Muscular Dystrophies; Low Back Pain
MeSH Terms: conditions — Multiple Sclerosis; Spinal Cord Injuries; Chronic Pain; Muscular Dystrophies; Low Back Pain

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- Pain Self-Management Arm #1 (Experimental): Pain Self-Management Intervention #1
  Interventions: Behavioral: Pain Self-Management Intervention #1
- Pain Self-Management Arm #2 (Experimental): Pain Self-Management Intervention #2
  Interventions: Behavioral: Pain Self-Management Intervention #2
- Pain Self-Management Arm #3 (Experimental): Pain Self-Management Intervention #3
  Interventions: Behavioral: Pain Self-Management Intervention #3
- Pain Self-Management Arm #4 (Experimental): Pain Self-Management Intervention #4
  Interventions: Behavioral: Pain Self-Management Intervention #4

INTERVENTIONS:
Behavioral: Pain Self-Management Intervention #1 — Pain Self-Management Intervention #1 will consist of four 60-minute sessions conducted in person over four weeks (1 session/week on average), scheduled at times convenient for participants (including evenings and weekends if necessary). The sessions will cover a variety of topics, including the definition of chronic pain, the physiological processes underlying chronic pain, common pain-related conditions such as sleep disturbance, and the effects of chronic pain. Participants will be encouraged to ask questions about and discuss the information presented during the treatment sessions.
  Arms: Pain Self-Management Arm #1
Behavioral: Pain Self-Management Intervention #2 — Pain Self-Management Intervention #2 will consist of four 60-minute sessions conducted in person over four weeks (1 session/week on average), scheduled at times convenient for participants (including evenings and weekends if necessary). Pain Self-Management Intervention #2 will emphasize cognitive restructuring skills to replace maladaptive pain-related thoughts with adaptive and reassuring ones. These skills include being able to: (1) develop awareness of one's thoughts; (2) identify and evaluate adaptive/helpful vs. unhelpful/maladaptive thoughts; and (3) develop alternative thoughts to maladaptive thoughts that are (a) realistic, (b) accurate, (c) reassuring, and (d) facilitate positive outcomes.
  Arms: Pain Self-Management Arm #2
Behavioral: Pain Self-Management Intervention #3 — Pain Self-Management Intervention #3 will consist of four 60-minute sessions conducted in person over four weeks (1 session/week on average), scheduled at times convenient for participants (including evenings and weekends if necessary). In Pain Self-Management Intervention #3, subjects will relax in a comfortable position with their eyes closed and simply listen to the clinician speak. The clinician will begin the session with a hypnotic induction focusing on being aware of sensations of relaxation, followed by suggestions for decreases in pain intensity and alterations in the sensory experience of "what are sometimes uncomfortable sensations" so that they are more comfortable.
  Arms: Pain Self-Management Arm #3
Behavioral: Pain Self-Management Intervention #4 — Pain Self-Management Intervention #4 will consist of four 60-minute sessions conducted in person over four weeks (1 session/week on average), scheduled at times convenient for participants (including evenings and weekends if necessary). Pain Self-Management Intervention #4 will use hypnotic strategies and suggestions for identifying adaptive cognitions and for making adaptive changes in cognitions more integrated into a participant's belief system.
  Arms: Pain Self-Management Arm #4

SUMMARY:
Many individuals with multiple sclerosis (MS), spinal cord injury (SCI), acquired amputation (AMP), muscular dystrophy (MD), and low back pain (LBP) experience pain. There has been little research on how to treat this pain. Different types of treatment that include self-hypnosis, education about chronic pain, and learning skills on how to change how a person thinks about his/her pain have been used to treat chronic pain in the general population. The purpose of this study is to see if these different treatments can help decrease pain in people with multiple sclerosis and spinal cord injury, and determine how and why these treatments are effective. A subject must have a diagnosis of MS,SCI, AMP, MD, or LBP, have chronic pain, and be at least 18 years old to participate.

DETAILED DESCRIPTION:
Individuals from the study's recruitment sources with the diagnoses listed above will be contacted by research staff via telephone and invited to be screened for participation. In addition, individuals interested in participating may contact research staff upon learning about the study through a description listed on an approved website or a referral. Research staff will use a recruitment script for purposes of screening subjects and explaining the study. In addition, the initial screening process will also include conducting a cognitive screening known as the 6-item cognitive screener.

Research staff will verify the diagnoses (MS, SCI, AMP, MD or LBP) of prospective subjects who have not been 'pre-verified' in one of three ways during the recruitment process:

1. Research staff will attempt to determine whether a subject from has a University of Washington Medical Center (UWMC)/Harborview Medical Center (HMC) medical record by conducting a simple search using a secure application.

   If research staff are unable to locate a medical record for the prospective subject from recruitment strategy #1, or if the individual is part of recruitment strategy #4 (i.e. if individual sees description of study on clinicaltrials.gov and contacts research staff), then one of two options will be pursued:
2. Subjects will be asked during the initial screening process if staff may review their medical records if they have received services at the UWMC/HMC since their diagnosis;
3. Subjects will be asked during the initial screening process if staff may contact a physician of their choice to verify their diagnosis if (a) they have not received services at the UWMC/HMC since their diagnosis; (b) they refuse to give staff permission to review their UWMC/HMC medical records; or (c) staff for some reason cannot find a UWMC/HMC medical record despite the subject attesting to being a patient at one time at the UWMC/HMC and giving staff permission to review his/her records.

Only individuals whose diagnosis has been verified (either via medical record review prior to/during screening or through verification via the subject's physician depending on recruitment source) will proceed with the psychological screening assessment.

Once a prospective subject has been screened and deemed eligible to participate, research staff will arrange a time and date for all subjects recruited into the study to participate in a telephone psychological screening assessment with one of the study's licensed clinicians (Drs. Jensen, Ehde, Molton, or Dillworth) or senior fellow (Elena Mendoza, a clinical psychologist). The study clinician will ask potential subjects some questions to assess the presence of active suicidal ideation or paranoid thoughts using an assessment sheet. Individuals who do have these types of thoughts will not be eligible for the study. Individuals will be referred to a mental health professional if he or she needs immediate attention.

Research staff will then arrange a time with the subject to attend in person what we call the initial intake session. At the beginning of the initial intake session, research staff will review a consent form with the subject and answer any questions he/she may have. The subject will complete and sign the consent form if he/she would like to participate. If the subject decides to enroll in the study, he/she will then be asked to complete a set of tasks testing memory and processing speed, participate in a relaxation and hypnotic exercise, and provide basic demographic information, as well as information about diagnosis and pain problem(s) he/she experiences. The initial intake session will last about 1.5 hours depending on the subject's answers.

The subject will then participate in a brain activity assessment at the Integrated Brain Imaging Center (IBIC) at the University of Washington that will take about one hour to complete. The brain activity assessment consists of an electroencephalogram (EEG), which measures the electrical activity in the brain through electrodes placed on the scalp. There is no risk of electrical shock. Research staff will place a damp electrode net on the subject's head that contains the electrodes that will measure the subject's brain activity. EEG activity will be collected with the subject's eyes closed. The research staff member will collect the data and ask the subject to remain as still as possible during the assessment. A research staff member will ask the subject his/her pain intensity during and after the assessment.

Subjects will be randomly assigned (by chance, like flipping a coin) to one of four treatment interventions. All four treatment interventions involve educating subjects about pain, discussing the impact of pain, and discussing different ways to manage it in hopes of decreasing subjects' pain and its impact on their lives. Two treatment interventions will also involve self-hypnosis. During self-hypnosis, subjects learn to enter a state of focused attention, and then change how they experience pain. All four treatment interventions are called "self-management" approaches to pain management. All of these treatments are commonly used in pain clinics and have been used to treat pain in persons with MS and SCI. We are interested in comparing the four different approaches to treating chronic pain.

A research staff member will also contact each subject six times by telephone during his/her participation in the study to complete three short interviews or assessments, 3-5 minutes long, and one longer assessment, about 30-40 minutes long, in a period of one week. These assessments will be completed one week prior to treatment, about halfway through the treatment period, after the completion of treatment, and 3-, 6- and 12-months after the subject completes treatment. The three shorter assessments will include questions about pain intensity. The fourth longer assessment will include questions about such things as how the subject thinks about pain, treatments for pain the subject has received, medications or drugs the subject has used, and any depressive symptoms the subject may have experienced.

We will also ask each subject to participate in a brain activity assessment following the end of treatment. The brain activity will be done the same way as described earlier and will take place at the Integrated Brain Imaging Center at the University of Washington.

ELIGIBILITY:
Inclusion Criteria:

1. 18 years of age or older;
2. diagnosis of SCI, MS, AMP, MD or LBP
3. moderate to severe chronic pain possibly related to MS, SCI, AMP, MD, or LBP that is persistent in nature;
4. able to read, speak, and understand English.

Exclusion Criteria:

1. severe cognitive impairment defined as two or more errors on the Six-Item Screen;
2. psychiatric condition or symptoms that would interfere with participation;
3. Pre-existing medical conditions that might interfere with EEG assessments.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 177 (Actual)
Dates: Start 2013-02 (Actual); Primary Completion 2018-01 (Actual); Study Completion 2018-01 (Actual)

PRIMARY OUTCOMES:
Change in average pain intensity pre-treatment to post-treatment | Pre-treatment, Mid-treatment, Post-treatment, 3-,6-, and 12 months following end of treatment.
  Average pain intensity will be assessed via telephone interviews using a 0-10 numerical rating scale (NRS) of average pain in the past 24 hours, four times within a 1-week period at each assessment point. The change in mean of these ratings will be used as the primary outcome measure of average daily pain intensity.

CONTACTS AND LOCATIONS:
Overall Officials: Mark Jensen, PhD, Principal Investigator — University of Washington
Locations (1):
- University of Washington, Ninth and Jefferson Building, Seattle, Washington, United States

REFERENCES:
- [Derived] de la Vega R, Sakulsriprasert P, Miro J, Jensen MP. Optimizing Pain Intensity Assessment in Clinical Trials: How Many Ratings are Needed to Best Balance the Need for Validity and to Minimize Assessment Burden? J Pain. 2024 Jul;25(7):104474. doi: 10.1016/j.jpain.2024.01.339. Epub 2024 Jan 15. PMID 38232864